CLINICAL TRIAL: NCT05403580
Title: Olanzapine for the Treatment of Chronic Nausea and/or Vomiting, Unrelated to Chemotherapy or Radiation, in Advanced Cancer Patients - A Confirmatory Phase III MNCCTN Trial
Brief Title: Olanzapine for the Treatment of Chronic Nausea and/or Vomiting in Patients With Advanced Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Closed due to slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MC211002; NCI-2022-02478 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC211002 (Other: Mayo Clinic in Rochester); 21-011317 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-05-19; First posted 2022-06-03 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (olanzapine) (Experimental): Patients receive olanzapine PO every night on days 1-28.
  Interventions: Drug: Olanzapine; Other: Questionnaire Administration
- Arm II (placebo, olanzapine) (Active Comparator): Patients receive placebo PO every night on days 1-2 and olanzapine PO every night on days 3-28.
  Interventions: Drug: Olanzapine; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Olanzapine — Given PO
  Other Names: LY 170053; Zyprexa; Zyprexa Zydis
Drug: Placebo Administration — Given PO
  Arms: Arm II (placebo, olanzapine)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares olanzapine to placebo in decreasing nausea and vomiting in patients with cancer that has spread to other places in the body (advanced). Patients with advanced cancer may experience nausea and/or vomiting that is unrelated to chemotherapy or radiation. Giving olanzapine may help reduce nausea and increase appetite in patients who have advanced cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To conduct a confirmatory phase III double-blind randomized clinical trial to evaluate the ability of olanzapine to decrease nausea in patients with advanced-cancer associated nausea/vomiting.

SECONDARY OBJECTIVES:

I. To evaluate toxicity associated with olanzapine in patients with advanced-cancer associated nausea/vomiting.

II. To evaluate the effect of olanzapine on appetite, vomiting, sedation, sleep, the use of other antiemetic agents, fatigue, and well-being.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive olanzapine orally (PO) every night on days 1-28.

ARM II: Patients receive placebo PO every night on days 1-2 and olanzapine PO every night on days 3-28.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histologically or cytologically-confirmed cancer in an advanced incurable stage
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Chronic nausea that has been present for at least one week (daily score > 5, on a 0-10 visual analogue scale)
* Serum creatinine < 2.0 mg/dl =< 120 days prior to registration
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) values < 3 times upper limits of normal =< 120 days prior to registration
* Negative pregnancy test done =< 14 days prior to registration, for persons of childbearing potential only
* Able to provide written informed consent
* Able to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

* Any of the following because this study involves: an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
* Received chemotherapy or radiation within the prior 14 days (advanced cancer patients receiving hormonal therapy or targeted therapy that does not come with a recommendation for prophylactic anti-emetic therapy are eligible)
* Receiving treatment with another antipsychotic agent such as risperidone, quetiapine, clozapine, phenothiazine or butyrophenone for =< 30 days prior to registration or planned during protocol therapy (patients may have received prochlorperazine and other phenothiazines as prior anti-emetic therapy)
* Those with concurrent use of ethyol; severe cognitive compromise; concurrent use of amifostine; concurrent use of quinolone antibiotic therapy; known hypersensitivity to olanzapine; or have planned chemotherapy or radiation during the 7 days following study initiation
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection (including human immunodeficiency virus [HIV])
  * Cardiac disease which, in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Inability to swallow oral formulations of the agent(s)
* Tube feeding or nasogastric tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in nausea score | Baseline to 24 hours of treatment
  Evaluated using Visual Analogue Scale. Nausea scores at baseline and after the first two days and the change scores, for the first 2 days, will be summarized using mean (standard deviation) and median (range). The change scores from baseline to the end of the first 2 days will be compared between arms using a two-sample t-test or a Wilcoxon rank sum test as appropriate. The difference in nausea change scores from baseline to 2 days post treatment initiation between the two arms will be estimated along with a 95% confidence interval.

SECONDARY OUTCOMES:
Daily nausea and vomiting scores | Up to 28 days
  Chronic nausea this is present for at least 1 week (worst daily nausea numeric rating scores needed to be greater than 3 on a 0-10 scale).
Daily episodes of vomiting/retching (number and time) | Up to 28 days
  Chronic nausea that is present for at least 1 week (worst daily nausea numeric rating scores needed to be greater than 3 on a 0-10 scale).
Utilization of rescue therapy | Up to 28 days
  Baseline evaluation that includes assessment of symptom intensity for appetite, nausea, fatigue, sedation, and pain, all measured and recorded on a numeric rating score. (0 indicated the worst possible; 10, best possible).
Incidence of adverse events with olanzapine | Up to 28 days
  Measured by patient reported outcome questionnaires and Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Charles L Loprinzi, Principal Investigator — Mayo Clinic in Rochester

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials